CLINICAL TRIAL: NCT05127174
Title: A Phase I/II Trial of Maintenance Fedratinib to Prevent Post-Transplant Relapse in Myeloproliferative Neoplasms
Brief Title: Maintenance Fedratinib to Prevent Post-Transplant Relapse in Myeloproliferative Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not advance to Phase 2
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20923; FEDR-CL-MF-PI-13906 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Myeloproliferative Neoplasm
Keywords: allogeneic hematopoietic cell transplant (HCT)
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Dose Level 1 (Experimental): Participants will take 200 mg fedratinib once daily by mouth.
  Interventions: Drug: Fedratinib Pill
- Phase 1: Dose Level 2 (Experimental): Participants will take 300 mg fedratinib once daily by mouth.
  Interventions: Drug: Fedratinib Pill
- Phase 1: Dose Level 3 (Experimental): Participants will take 400 mg fedratinib once daily by mouth.
  Interventions: Drug: Fedratinib Pill
- Phase 2: Treatment at Recommended Phase 2 Dose (RP2D) (Experimental): Participants will take fedratinib at the dose determined in the phase 1 portion of this study, once daily by mouth.
  Interventions: Drug: Fedratinib Pill

INTERVENTIONS:
Drug: Fedratinib Pill — Fedratinib is taken orally once per day, in 100 mg capsules. Fedratinib is an oral kinase inhibitor with activity against wild type and mutationally activated Janus Associated Kinase 2 (JAK2) and FMS-like tyrosine kinase 3 (FLT3).
  Other Names: Inrebic

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of fedratinib as maintenance therapy in participants with myeloproliferative neoplasms (MPNs) after allogeneic hematopoietic cell transplant (HCT).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the informed consent form (ICF)
* Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) of 0, 1 or 2
* Must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
* Willing and able to adhere to the study visit schedule and other protocol requirements.
* Philadelphia chromosome negative myeloproliferative disease (including polycythemia vera, myelofibrosis, and essential thrombocytosis, chronic myelomonocytic leukemia, atypical chronic myelogenous leukemia, myelodysplastic syndrome/myeloproliferative neoplasm-unclassified, MPN not otherwise specified) having undergone first allogeneic HCT.
* Engraftment including >95% myeloid cell donor chimerism and Absolute neutrophil count (ANC) > 1.0 x 109/L
* Platelets > 50 x 109/L with no platelet transfusions in the prior 7 days
* Absence of disease progression as defined by International Working Group (IWG) Myeloproliferative Neoplasm Response Criteria
* Acute GVHD of the skin is permitted if prednisone has been tapered to <0.25 mg/kg with continued response
* Females of childbearing potential (FCBP) must:

  1. Have a negative pregnancy tests as verified by the Investigator during screening prior to enrollment (a second pregnancy test will be collected prior to therapy as below). She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.
  2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use and be able to comply with highly effective contraception** without interruption, -14 days prior to starting investigational product, during the study treatment (including dose interruptions), and for 30 days after discontinuation of study treatment.

Note: A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

* Male participants must:

Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 30 days following investigational product discontinuation, or longer if required for each compound and/or by local regulations, even if he has undergone a successful vasectomy.

* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

** Agreement to use highly effective methods of contraception that alone or in combination resulting in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly throughout the course of the study. Such methods include: Combined (estrogen and progestogen containing) hormonal contraception: Oral; Intravaginal; Transdermal; Progestogen-only hormonal contraception associated with inhibition of ovulation: Oral; Injectable hormonal contraception; Implantable hormonal contraception; Placement of an intrauterine device; Placement of an intrauterine hormone-releasing system; Bilateral tubal occlusion; Vasectomized partner.

Exclusion Criteria:

* Acute GVHD of the gut or liver currently on systemic therapy. Patients who have completed systemic therapy and are asymptomatic may be enrolled.
* Treatment with JAK2 inhibitor within 14 days prior to enrollment.
* Any of the laboratory abnormalities outlined in protocol
* Pregnant or lactating female
* Prior history of Wernicke's encephalopathy (WE)
* Has signs or symptoms of encephalopathy, including Wernicke's Encephalopathy (e.g. severe ataxia, ocular paralysis or cerebellar signs) in which case thiamine deficiency needs to be excluded and a brain MRI might be required to exclude possible Wernicke's encephalopathy
* Patient with concomitant treatment with or use of pharmaceutical or herbal agents known to be strong inducers of CYP3A4. However, if a patient is started on a strong CYP3A4 inducer while on fedratinib, the dose must be adjusted as described in the drug-drug interaction section below.
* Thiamine levels below the normal range, per institutional standard, may enroll but must be corrected to the normal range before initiating treatment with fedratinib (See section 6.5.1). Normalized thiamine level must be confirmed within 10 days of starting fedratinib therapy.
* On any chemotherapy, immunomodulatory drug therapy (e.g., thalidomide, interferon-alpha), Anagrelide, or concurrent JAK2 inhibitor. Patients who have had exposure to hydroxyurea (e.g., hydrea) in the past may be enrolled into the study as long as it has not been administered within 14 days prior to initiation of fedratinib
* On treatment with myeloid growth (e.g. G-CSF) factor within 14 days prior to initiation of fedratinib
* On treatment with aspirin with doses > 150 mg daily
* Major surgery within 28 days before starting fedratinib
* Diagnosis of chronic liver disease (e.g., chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemochromatosis, non-alcoholic steatohepatitis
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4)
* Known human immunodeficiency virus (HIV), evidence of active infectious Hepatitis B (Hep B), and/or evidence of active Hepatitis C (Hep C)
* Serious active infection
* Presence of any significant gastric or other disorder that would inhibit absorption of oral medication
* Concurrent active malignancy requiring therapy. Localized skin basal cell or squamous cell carcinomas are permitted.
* Bone marrow blast percentage greater than 10%.
* Unable to swallow capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Phase 1: Recommended Phase 2 Dose | Up to 1 year
  Participants will be treated at increasing dose levels to determine the Recommended Phase 2 Dose (RP2D). The RP2D will be defined as the highest dose level with a true dose limiting toxicity (DLT) rate <33%.
Phase 2: Progression Free Survival | at 1 year
  Progression Free Survival defined as the time from start of treatment to the time of disease progression or death.

SECONDARY OUTCOMES:
Number of Participants who develop Chronic Graft vs Host Disease | 1 year
  Number of Participants who develop Chronic Graft vs Host Disease (GVHD)
Overall Survival | 1 year
  Overall Survival (OS) is defined as the time from the date of HCT (Hematopoietic Cell Transplant) to the date of death due to any cause.
Relapse Rate | 1 year
  Disease relapse rate, defined as the incidence of signs of symptoms of disease returning after a period of improvement.
Transplant related mortality rate | 1 year
  Rate of deaths related to Hematopoietic Cell Transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Taiga Nishihori, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No